CLINICAL TRIAL: NCT01828515
Title: Vilazodone for Corticosteroid-Induced Memory Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Sherwood Brown, MD, PhD, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 082012-082
Record Dates: First submitted 2012-11-07; First posted 2013-04-10 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Memory Impairment
MeSH Terms: conditions — Memory Disorders | interventions — Vilazodone Hydrochloride; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vilazodone and Hydrocortisone, then Placebo and Hydrocortisone (Experimental): Vilazodone titrated to 10 mg x 7 days, 20 mg x 7 days and 40 mg x 5 days (19 days) and hydrocortisone 160 mg x 4 days (days 16-19) following vilazodone pre-treatment. After a 23 day medication washout the procedure will be repeated using placebo daily for 19 days and hydrocortisone 160 mg x 4 days (days 16-19) following placebo pre-treatment.
  Interventions: Drug: Vilazodone; Drug: Placebo; Drug: Hydrocortisone
- Placebo and Hydrocortisone, then Vilazodone and Hydrocortisone (Experimental): Placebo daily for 19 days and hydrocortisone 160 mg x 4 days (days 16-19) following placebo pre-treatment. After a 23 day medication washout the procedure will be repeated using Vilazodone titrated to 10 mg x 7 days, 20 mg x 7 days and 40 mg x 5 days (19 days) and hydrocortisone 160 mg x 4 days (days 16-19) following vilazodone pre-treatment.
  Interventions: Drug: Vilazodone; Drug: Placebo; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Vilazodone — Participants will be randomized to either vilazodone or placebo titrated as follows: 10 mg x 7 days, 20 mg x 7 days and 40 mg x 5 days.
  Other Names: Viibryd
Drug: Placebo
Drug: Hydrocortisone — Participants receive 160 mg x 4 days after vilazodone or placebo pre-treatment

SUMMARY:
The purpose of this study is to examine whether vilazodone attenuates the memory and mood effects of corticosteroids on the human hippocampus in 24 healthy controls.

DETAILED DESCRIPTION:
In animals and humans, stress and corticosteroid excess are associated with changes in hippocampal structure and functioning. These findings have important implications to the millions of patients taking prescription corticosteroids and to patients with major depressive disorder or bipolar disorder who have elevated cortisol levels and memory impairment. The investigators believe that vilazodone may be a medication that can block the effects of hydrocortisone on the human hippocampus. The investigators propose to examine whether vilazodone attenuates the effects of corticosteroids in a randomized, double-blind, placebo-controlled pilot study using a within-subject crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women age 18-50 years
* Education of ≥ 12 years and baseline RAVLT total words recalled score ≥ 35 (normal baseline memory)
* BMI between 18.5-30 (not underweight or obese)

Exclusion Criteria:

* History of major psychiatric illness defined as major depressive disorder, bipolar disorder, posttraumatic stress disorder, panic disorder, schizoaffective disorder, schizophrenia, eating disorders, or drug/alcohol abuse/dependence or current tobacco use
* History of neurological disorders including seizures, brain surgery, multiple sclerosis, Parkinson's disease
* Taking CNS-acting medications within 30 days of study
* History of allergic reaction or medical contraindication to vilazodone or hydrocortisone
* Significant medical conditions (e.g., myocardial infarction, cancer, diabetes)
* Vulnerable population including pregnant or nursing women, the incarcerated, and severe cognitive disorders
* Baseline HRSD (Hamilton Rating Scale for Depression) > 7 or current suicidal ideation or history of suicide attempt
* History of systemic Corticosteroid (CS) use or recent (past 6 months) inhaled CS use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, M.D., Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 participants with at least one post-baseline visit were recruited at our research clinic in Dallas, TX and included for analysis.
Pre-assignment Details: Healthy control participants without any history of major psychiatric illness, drug/alcohol abuse/dependence, history of neurological disorders, or significant medical conditions were included.
Groups:
- Vilazodone and Hydrocortisone,Then Placebo and Hydrocortisone: Vilazodone was initiated at 10 mg/day for 7 days and increased to 20 mg/day for 7 days. After that time an additional increase to 40 mg/day for 5 days (totaling 19 days). On the 2nd day of the 40 mg a day portion, 160 mg of hydrocortisone/day was given for 4 days. After a washout period of 23 days, placebo was given for 19 days and hydrocortisone was given for 4 days.
- Placebo and Hydrocortisone, Then Vilazodone and Hydrocortisone: Placebo was given for 19 days and hydrocortisone was given for 4 days. After a washout period of 23 days, Vilazodone was initiated at 10 mg/day for 7 days and increased to 20 mg/day for 7 days. After that time an additional increase to 40 mg/day for 5 days (totaling 19 days). On the 2nd day of the 40 mg a day portion, 160 mg of hydrocortisone/day was given for 4 days.
Period: First Intervention (19 Days)
Arm/Group | Vilazodone and Hydrocortisone,Then Placebo and Hydrocortisone | Placebo and Hydrocortisone, Then Vilazodone and Hydrocortisone
Started | 13 | 11
Completed | 11 | 9
Not Completed | 2 | 2
Period: Washout (23 Days)
Arm/Group | Vilazodone and Hydrocortisone,Then Placebo and Hydrocortisone | Placebo and Hydrocortisone, Then Vilazodone and Hydrocortisone
Started | 11 | 9
Completed | 6 | 8
Not Completed | 5 | 1
Period: Second Intervention (19 Days)
Arm/Group | Vilazodone and Hydrocortisone,Then Placebo and Hydrocortisone | Placebo and Hydrocortisone, Then Vilazodone and Hydrocortisone
Started | 6 | 8
Completed | 6 | 5
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Vilazodone and hydrocortisone or placebo and hydrocortisone.
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline RAVLT (Rey Auditory Verbal Learning Test) Total T-Score at Day 19
Description: The Rey Auditory Verbal Learning Test (RAVLT) measures verbal or declarative learning and memory. The test consists of 15 nouns read aloud for five consecutive trials with each trial followed by a free-recall trial. Following the fifth trial, an interference list of 15 different words is presented followed by a free-recall trial of that list. Delayed recall of the first list is tested immediately following the interference list and after a 20-minute delay. Equivalent, alternative versions (different words) were used to minimize practice or learning effects from repeated administration. The raw scores (number of words correct across trials 1-5) are converted to standardized T-scores (M=50; SD=10). This score is used to determine the participant's performance in relation to norm-referenced expectations based on age and sex. Higher score reflects better performance, and the values reflect scores at baseline minus the scores at Day 19.
Time Frame: Baseline and Day 19
Population: All participants who received at least one dose of each intervention and completed all study visits were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Vilazodone and Hydrocortisone: Vilazodone was initiated at 10 mg/day for 7 days and increased to 20 mg/day for 7 days. After that time an additional increase to 40 mg/day for 5 days (totaling 19 days). On the 2nd day of the 40 mg a day portion, 160 mg of hydrocortisone/day was given for 4 days.
- Placebo and Hydrocortisone: Placebo was given for 19 days and hydrocortisone was given for 4 days.
Arm/Group | Vilazodone and Hydrocortisone | Placebo and Hydrocortisone
Number analyzed (Participants) | 14 | 14
T-score | -3 (12.48) | 0 (7.98)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study between baseline and end of study procedures (after 2 complete cycles of treatment) or an average of 2 months.
Description: Adverse events were assessed by a weekly questionnaire at each appointment.
Groups:
- Vilazodone and Hydrocortisone: Vilazodone was initiated at 10 mg/day for 7 days and increased to 20 mg/day for 7 days. After that time an additional increase to 40 mg/day for 5 days (totaling 19 days).
- Placebo and Hydrocortisone: Placebo group received medication in identical color/sizes as the Vilazodone group. Placebo was given for 19 days.
Arm/Group | Vilazodone and Hydrocortisone | Placebo and Hydrocortisone
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 2/24 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vilazodone and Hydrocortisone (N=24) | Placebo and Hydrocortisone (N=24)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not related to the medication or study
Varicocele (Vascular disorders) | 1 (1) | 0 (0) — Not related to the medication or study

LIMITATIONS AND CAVEATS:
The sample size was modest and attrition rate was high; The study also lacked neuroimaging or other biomarkers to correlate changes in memory; Study drug adherence was only assessed with pill counts not with metered dosing counts or blood levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less